CLINICAL TRIAL: NCT03642080
Title: Imaging Biomarkers to Predict Responsiveness to Tumor Treating Fields in Patients With High Grade Glioma
Brief Title: MRI Predictors of Response to Tumor Treating Fields
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Theodore Yanagihara, Assistant Professor of Clinical Radiation Oncology, New York Presbyterian Brooklyn Methodist Hospital
Other Study IDs: 1137708
Record Dates: First submitted 2018-04-13; First posted 2018-08-22 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Glioblastoma: Patients with a diagnosis of newly diagnosed or recurrent glioblastoma who have been treated with radiation and temozolomide and are being offered tumor treated fields.

SUMMARY:
Patients with glioblastoma, an aggressive brain tumor, are recommended to undergo treatment with tumor treating fields using the Optune device as part of standard of care therapy. While undergoing treatment, patients are monitored regularly with brain MRI scans to look for tumor progression, but there are currently no means to predict which, or when, patients will progress. The purpose of the current study is to prospectively analyze these MRI scans to look for subtle imaging markers that can predict for future brain tumor progression while undergoing tumor treating field therapy.

DETAILED DESCRIPTION:
The proposed trial involves the prospective collection of imaging data at standard clinical time points before and during treatment with TTFields. All patients who are offered treatment with TTFields will also be offered enrollment in this non-randomized, observational study. Imaging data will include the standard battery of MRI sequences, which includes DWI and ADC reconstruction. These data will be collected at standard time points and the proposed study will not rely on any additional imaging or tests outside of the clinical standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18 or older with newly diagnosed WHO grade IV glioblastoma or patients with recurrent glioblastoma not previously treated with TTFields.
* Patients may have undergone surgical resection or biopsy.
* Residual tumor, absence of treatment with temozolomide or radiation therapy will not be an exclusion criteria for the study.

Exclusion Criteria:

* Patients previously treated with TTFields will not be included in the study.
* Patients will also be excluded if they are undergoing active treatment with systemic agents, including bevacizumab, during treatment with TTFields.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient with newly diagnosed or with recurrent glioblastoma who meet the eligibility criteria of the study.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression of disease | Until discontinuation of tumor treating fields, progression or death. This will be evaluated by imaging and clinical exam from the time of trial enrollment until up to 36 months at approximately three-month intervals.
  Clinical or radiographic disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Adel Guirguis, MD, MS, Study Director — New York Presbyterian Hospital - Brooklyn Methodist Hospital
Locations (1):
- New York Presbyterian - Brooklyn Methodist Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided